CLINICAL TRIAL: NCT04333173
Title: ENDOVASCULAR THERAPY REGISTRY FOR ERECTILE DYSFUNCTION
Brief Title: Endovascular Therapy for Erectile Dysfunction
Acronym: RE-ACTION
Status: Completed | Type: Observational
Sponsor: Clinica San Gaudenzio (Other)
Responsible Party: Principal Investigator, Giuseppe Sangiorgi, Prof, Clinica San Gaudenzio
Other Study IDs: 101010
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Erectile Dysfunction
Keywords: ED
MeSH Terms: conditions — Erectile Dysfunction | interventions — Endovascular Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Active endovascular treatment: Patients with erectile dysfunction (ED) and no-response to phosphodiesterase-5 inhibitors for at least 6 months before enrollment
  Interventions: Procedure: endovascular procedure

INTERVENTIONS:
Procedure: endovascular procedure — Endovascular therapies for erectile dysfunction

SUMMARY:
Brief Summary: Background and pathophysiology Erectile dysfunction is a serious disease with a significant impact on the quality of life. Male erection is a complex mechanism that involves neuro-vascular tissue responses with several phases including arterial dilatation, smooth muscle cells relaxation and ultimately veno-occlusive activation. Vasculogenic erectile dysfunction can be divided in arteriogenic (when there is insufficiency of arterial component of erection due to atherosclerotic plaque encroachment of the penile arteries) or venogenic (where there is insufficiency of the venous component of erection for venous endoleak) Standard treatment Erectile dysfunction is commonly treated by oral phosphodiesterase-5-inhbitor (PDE5i) administration. However, up to 50% of men have a suboptimal response to PDE5-i therapy with the need of additional therapies. New treatment Only recently several studies have been published on percutaneous treatment of ED using POBA, Drug eluting balloons (both paclitaxel and sirolimus, PEB and SES) and drug eluting stents (DES).

Aim of the study The study was aimed at evaluating both arteriogenic and venogenic endovascular treatments in patients affected by erectile dysfunction in an Italian patient cohort.

DETAILED DESCRIPTION:
Detailed Description: The objective of this study is to evaluate of the safety and feasibility of endovascular therapies in segmental atherosclerotic lesions of the internal pudendal arteries among men with erectile dysfunction (ED) and no-response to phosphodiesterase-5 inhibitors for at least 6 months either at increasing dosage or with different drugs routinely utilized in this setting) before enrollment. All patients will be screened by IIEF-5 questionnaire (IEF-5 Score < 15 points); Penile Dynamic Doppler ultrasound with intracavernous injection of Caverject (cut-off for Inflow insufficiency: PSV <25 cm s-1, EDV <5 cm s-1, RI > 0.8; cut-off for Venous leakage: PSV > 25 cm s-1, EDV > 5 cm s-1, RI < 0.8; cut-off for mixed pathology: PSV < 25 cm s-1, EDV > 5 cm s-1, RI < 0.8); and/or positive angio-CT scan for stenosis of the penile arteries of venous insufficiency. All patients will be treated either by POBA+PES/SES or in case of suboptimal result (angiographic residual stenosis > 30%) with DES implantation. All patients will be discharged with dual antiplatelet therapy for 3 months and with Cialis 5 mg daily for 30 days. Patients will be followed at 1 mos with IIEF questionnaire, 3 months with IIE-5 questionnaire, 8 months with IIEF questionnaire and Dynamic Doppler ultrasound evaluation, and 12 months with IIEF-5 questionnaire and Dynamic Doppler ultrasound evaluation. Primary endpoints will be the delta of IEF-5 score between basal and 8 months FU (>5 points). Delta PSV (>8 points of cm/sec at the Dynamic Doppler evaluation) between basal and 8 mos follow-up. 1. Secondary endpoints will be a) Incidence of MAE (Death, MI, Stroke), 2) Binary restenosis and late loss in patients who will repeat control angiography if clinically indicated for ED recurrence (clinically evaluated by either needs to reintroduce/increase PDEF5i dosage on-demand, delta IEF-5 <5 compared to 1 mos FU after 6 mos FU) or in patients with bilateral disease with scheduled procedure after 6 mos FU from the index procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Be able to understand and sign a witnessed informed consent for the procedure
* Eligibility for percutaneous peripheral intervention
* Baseline IIEF-5 score evaluation < 15
* PSV < 25 cm/sec
* Stable hemodynamic conditions
* Normal ejection fraction
* Being refractory to oral PDE5-I for at least 6 months before enrollement
* Treatable angiographic lesions of the pudendal arteries

Exclusion Criteria:

* Heart failure
* Hemodynamic instability
* Basal IIEF-5 and doppler examination
* Blood count not within normal ranges
* No history of bleeding or coagulopathy
* No other serious medical illness
* Other investigational drug or device study
* Pudendal artery < 1.5 mm and lesion lenght greater than 80 mm by visual estimation
* Pudendal restenosis from previous intervention

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Patients with erectile dysfunction (ED) and no-response to phosphodiesterase-5 inhibitors for at least 6 months before enrollment
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
IEF-5 SCORE VARIATION AFTER ENDOVASCULAR | 6 months
  INTERNATIONAL INDEX OF ERECTILE FUNCTION

SECONDARY OUTCOMES:
PSV VARIATION AFTER ENDOVASCULAR TREATMENT | 6 month
  PUDENDAL DOPPLER PEAK SYSTOLIC VELOCITY
ADVERSE EVENTS | 6-12 months
  Procedural complications; cardiovascular events during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Cuore, Novara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sangiorgi G, Colantonio R, Antonini G, Savino A, Sperandio M. [Percutaneous intervention therapy for vascular erectile dysfunction]. G Ital Cardiol (Rome). 2016 Oct;17(10 Suppl 1):12S-21. doi: 10.1714/2372.25474. Italian. PMID 27729664
- [Background] Doppalapudi SK, Wajswol E, Shukla PA, Kolber MK, Singh MK, Kumar A, Fischman A, Rastinehad AR. Endovascular Therapy for Vasculogenic Erectile Dysfunction: A Systematic Review and Meta-Analysis of Arterial and Venous Therapies. J Vasc Interv Radiol. 2019 Aug;30(8):1251-1258.e2. doi: 10.1016/j.jvir.2019.01.024. Epub 2019 May 17. PMID 31104902
- [Background] Diehm N, Marggi S, Ueki Y, Schumacher D, Keo HH, Regli C, Do DD, Moeltgen T, Grimsehl P, Wyler S, Schoenhofen H, Raber L, Schumacher M. Endovascular Therapy for Erectile Dysfunction-Who Benefits Most? Insights From a Single-Center Experience. J Endovasc Ther. 2019 Apr;26(2):181-190. doi: 10.1177/1526602819829903. Epub 2019 Feb 11. PMID 30741067